CLINICAL TRIAL: NCT04203732
Title: Evaluation of Anesthetic Techniques in Outpatient Total Joint Replacement Surgery in an Integrated Health Care Delivery System
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 1502384-1
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Anesthesia Morbidity; Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Retrospective Cohort; Anesthetic Technique; Total Joint Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Joint Arthroplasty: The cohort includes patients undergoing outpatient primary total joint replacement surgeries from 2017 to 2019. Primary total joint surgery is defined as patients who undergo unilateral total knee replacement or total hip replacement for the first time during the study years
  Interventions: Procedure: Anesthesia Type

INTERVENTIONS:
Procedure: Anesthesia Type — The anesthetic type either general anesthesia or neuraxial anesthesia is the intervention type for patients undergoing primary total joint arthroplasty of the knee or hip.
  Other Names: Anesthetic Technique

SUMMARY:
The study is a retrospective cohort study of adult patients undergoing outpatient primary unilateral total knee or total hip replacement surgeries from 2017 to 2019 assessing for difference in anesthetic techniques and outcomes.

DETAILED DESCRIPTION:
The study is a retrospective cohort study of adult patients undergoing outpatient primary unilateral total knee or total hip replacement surgeries from 2017 to 2019. The purpose of the study is to evaluate the effects of anesthetic techniques for primary total joint replacement in Northern California Kaiser Permanente. The primary objective is to determine if there are clinically and statistically significant differences between the outcomes of general anesthesia and neuraxial anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 - IV patients
* Age > 18
* Primary total hip/knee replacement

Exclusion Criteria:

* Total joint replacement for oncologic tumors
* Emergent surgery
* Age < 17
* Pregnant Female
* Neuraxial anesthesia conversion to general anesthesia
* Revision total joint replacement
* Bilateral total joint replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary total joint surgery patients who undergo unilateral total knee replacement or total hip replacement for the first time during the study years of 2017 to 2019.
Sampling Method: Non-Probability Sample
Enrollment: 12466 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Morbidity | 30-day postoperative
  30-day Postoperative Morbidity including surgical site infection (defined as infection involving the skin or subcutaneous tissue of the incision, deep incisional infection defined as infected tissue below the subcutaneous tissue including fascia and muscle), major coronary events (defined as nonfatal myocardial infarction, heart failure, ventricular tachycardia, cardiac arrest), pneumonia, urinary tract infection, venous thromboembolism, pulmonary embolism, cerebrovascular accident, renal injury/failure (Defined as increase in baseline creatinine 2 fold/3fold respectively).

SECONDARY OUTCOMES:
Postoperative Mortality | 30-day postoperative
  30-day postoperative mortality - all cause
Postoperative readmission | 30-day postoperative
  30-day postoperative readmission - all cause
Intraoperative blood loss and transfusion rates | Day of surgery
  Measurement of blood loss by mL recorded on record. Measurement of packed red blood cells transfused by unit pack.
Intraoperative opioid use | Day of surgery
  Defined by type of analgesic medication and total morphine equivalence
Postoperative opioid use | Day of surgery
  Defined by type of analgesic medication and total morphine equivalence
Postoperative Pain Scores | Day of surgery
  Numerical Rating Scale of postsurgical pain measured until discharge from hospital. Numerical rating scale for pain is described as a scale from a minimum of 0, associated with no pain, to a maximum of 10, associated with the worst possible pain. A higher number is associated with a worse outcome.
Postoperative nausea and vomiting | Day of surgery
  Rate of PONV after surgery
Length of postsurgical hospital stay | Day of surgery
  Length of time defined from end of intraoperative time to discharge from hospital time

CONTACTS AND LOCATIONS:
Overall Officials: Edward N Yap, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, South San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu VX, Rosas E, Hwang J, Cain E, Foss-Durant A, Clopp M, Huang M, Lee DC, Mustille A, Kipnis P, Parodi S. Enhanced Recovery After Surgery Program Implementation in 2 Surgical Populations in an Integrated Health Care Delivery System. JAMA Surg. 2017 Jul 19;152(7):e171032. doi: 10.1001/jamasurg.2017.1032. Epub 2017 Jul 19. PMID 28492816
- [Background] Berger RA, Sanders SA, Thill ES, Sporer SM, Della Valle C. Newer anesthesia and rehabilitation protocols enable outpatient hip replacement in selected patients. Clin Orthop Relat Res. 2009 Jun;467(6):1424-30. doi: 10.1007/s11999-009-0741-x. Epub 2009 Feb 28. PMID 19252961
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Holte K, Kehlet H. Epidural anaesthesia and analgesia - effects on surgical stress responses and implications for postoperative nutrition. Clin Nutr. 2002 Jun;21(3):199-206. doi: 10.1054/clnu.2001.0514. PMID 12127927
- [Background] Hu S, Zhang ZY, Hua YQ, Li J, Cai ZD. A comparison of regional and general anaesthesia for total replacement of the hip or knee: a meta-analysis. J Bone Joint Surg Br. 2009 Jul;91(7):935-42. doi: 10.1302/0301-620X.91B7.21538. PMID 19567860
- [Background] Memtsoudis SG, Sun X, Chiu YL, Stundner O, Liu SS, Banerjee S, Mazumdar M, Sharrock NE. Perioperative comparative effectiveness of anesthetic technique in orthopedic patients. Anesthesiology. 2013 May;118(5):1046-58. doi: 10.1097/ALN.0b013e318286061d. PMID 23612126
- [Background] Pugely AJ, Martin CT, Gao Y, Mendoza-Lattes S, Callaghan JJ. Differences in short-term complications between spinal and general anesthesia for primary total knee arthroplasty. J Bone Joint Surg Am. 2013 Feb 6;95(3):193-9. doi: 10.2106/JBJS.K.01682. PMID 23269359
- [Background] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Background] Macfarlane AJ, Prasad GA, Chan VW, Brull R. Does regional anaesthesia improve outcome after total hip arthroplasty? A systematic review. Br J Anaesth. 2009 Sep;103(3):335-45. doi: 10.1093/bja/aep208. Epub 2009 Jul 23. PMID 19628483
- [Background] Kehlet H, Aasvang EK. Regional or general anesthesia for fast-track hip and knee replacement - what is the evidence? F1000Res. 2015 Dec 15;4:F1000 Faculty Rev-1449. doi: 10.12688/f1000research.7100.1. eCollection 2015. PMID 26918127
- [Background] Harsten A, Kehlet H, Toksvig-Larsen S. Recovery after total intravenous general anaesthesia or spinal anaesthesia for total knee arthroplasty: a randomized trial. Br J Anaesth. 2013 Sep;111(3):391-9. doi: 10.1093/bja/aet104. Epub 2013 Apr 11. PMID 23578860
- [Background] Harsten A, Kehlet H, Ljung P, Toksvig-Larsen S. Total intravenous general anaesthesia vs. spinal anaesthesia for total hip arthroplasty: a randomised, controlled trial. Acta Anaesthesiol Scand. 2015 Mar;59(3):298-309. doi: 10.1111/aas.12456. Epub 2014 Dec 18. PMID 25522681
- [Background] Deyo RA, Cherkin DC, Ciol MA. Adapting a clinical comorbidity index for use with ICD-9-CM administrative databases. J Clin Epidemiol. 1992 Jun;45(6):613-9. doi: 10.1016/0895-4356(92)90133-8. PMID 1607900
- [Derived] Yap E, Wei J, Webb C, Ng K, Behrends M. Neuraxial and general anesthesia for outpatient total joint arthroplasty result in similarly low rates of major perioperative complications: a multicentered cohort study. Reg Anesth Pain Med. 2022 May;47(5):294-300. doi: 10.1136/rapm-2021-103189. Epub 2022 Jan 6. PMID 34992150